CLINICAL TRIAL: NCT00413439
Title: Open Label, Multi-center, Sequential Group Clinical Study to Determine the Safety and Efficacy of Escalating Dosing Regimens of Intravenous BAL8557 in the Prophylaxis of Patients Undergoing Chemotherapy for Acute Myeloid Leukemia
Brief Title: Safety, Efficacy and Pharmacokinetics of an Antifungal in Patients Undergoing Chemotherapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WSA-CS-002; 2005-005294-30 (EudraCT Number)
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Isavuconazole; BAL8557; ASP9766; chemotherapy; prophylaxis; systemic fungal infection
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose isavuconazole intravenous solution (Experimental)
  Interventions: Drug: Isavuconazole
- High dose isavuconazole intravenous solution or oral capsules (Experimental)
  Interventions: Drug: Isavuconazole

INTERVENTIONS:
Drug: Isavuconazole — Intravenous solution or oral capsules
  Other Names: ASP9766; BAL8557

SUMMARY:
Patients who undergo chemotherapy for leukemia will receive study medication for prevention of fungal infections. The study investigates the safety and tolerability of two different dosages, the efficacy in prevention of fungal diseases.

DETAILED DESCRIPTION:
Patients with Acute Myeloid Leukemia who undergo aggressive chemotherapy are due to immunosuppression susceptible to infections, including fungal infections. As the failure rate in the treatment of invasive fungal infections is high, prophylaxis is frequently recommended. This open label study investigates the safety and tolerability of two different dosages of a water soluble azole antifungal, as well as the efficacy in prevention of invasive fungal infections and pharmacokinetic data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute myeloid leukemia
* patients entering first induction treatment; or subsequent chemotherapy if no prior invasive fungal infection was observed
* expected to be neutropenic for >9 and <28 days after enrollment
* women of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

* patients who received any systemic antifungal therapy for more than 72 hours prior to first administration of study medication. Topical polyenes or nystatin are acceptable but should be discontinued during the study
* patients who received systemic antifungal therapy for proven or probable fungal infection in the last 12 months
* patients with fever defined as central body temperature of > 38°C
* known hypersensitivity to azoles or any component of the study medication
* concomitant use of rifampicin, rifabutin, ergots alkaloids, terfenadine, astemizole, cisapride, pimozide, quinidine, long acting barbiturates, neostigmine, and carbamazepine
* hepatic or severe renal dysfunction
* patients with a medical history of oliguria unresponsive to fluid challenge
* patients with a concomitant medical condition that may be an unacceptable additional risk to the patient should he/she participate in the study
* treatment with any investigational drug within 30 days prior to the first administration of study medication except open label chemotherapy protocols
* suspected other or additional cause for neutropenia or immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the recording of adverse events, laboratory tests, and electrocardiograms (ECGs) | Up to Day 28

SECONDARY OUTCOMES:
Efficacy assessed by the frequency of invasive fungal infections | Up to Day 28
Pharmacokinetics: drug plasma levels | Up to Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cornely, MD, Principal Investigator — University of Cologne
Locations (4):
- Germany (4):
  - Bremen
  - University Cologne, Cologne
  - Frankfurt
  - Mainz

REFERENCES:
- [Derived] Cornely OA, Bohme A, Schmitt-Hoffmann A, Ullmann AJ. Safety and pharmacokinetics of isavuconazole as antifungal prophylaxis in acute myeloid leukemia patients with neutropenia: results of a phase 2, dose escalation study. Antimicrob Agents Chemother. 2015 Apr;59(4):2078-85. doi: 10.1128/AAC.04569-14. Epub 2015 Jan 26. PMID 25624327